CLINICAL TRIAL: NCT01611207
Title: Randomised Controlled Study to Evaluate the Efficacy of the Treatment of Iatrogenic Subcutaneous Abdominal Wounds (ISAW) After Surgery by Application of Negative Pressure Wound Therapy (NPWT) in Comparison to Standard Conventional Wound Therapy (SCWT) of the Clinical Routine.
Brief Title: Evaluate the Efficacy of the Treatment of Iatrogenic Subcutaneous Abdominal Wounds (ISAW) After Surgery by Application of Negative Pressure Wound Therapy (NPWT) in Comparison to Standard Conventional Wound Therapy (SCWT) of the Clinical Routine
Acronym: ISAW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient recruitment was behind target, no successful completion of the planned patient numbers within trial period could be expected
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Kinetic Concepts, Inc. (Industry); Smith & Nephew Wound Management Inc (Industry)
Responsible Party: Principal Investigator, Dr. Marcus Redaèlli, Administative and scientific head of staffed offices of Interdisciplinary Centre for Health Services Research, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-2012; DRKS ID 00003498 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2012-03-28; First posted 2012-06-04 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Abdominal Wounds; Wound-healing Impairments
Keywords: wound healing impairments,; negative pressure wound therapy,; health services research,; germany
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): Used therapy systems
  Interventions: Device: Negative Pressure Wound Therapy
- Standard Conventional Wound Therapy (Active Comparator): Standard conventional wound therapy according to current evidence-based guideline (basic and advanced methods of wound treatment)
  Interventions: Other: Standard Wound Therapy

INTERVENTIONS:
Device: Negative Pressure Wound Therapy — KCI. V.A.C. Freedom; Acti V.A.C.; INFO V.A.C. to be used with the V.A.C. Granufoam (black), V.A.C. Granufoam Silver and V.A.C. WhiteFoam Smith & Nephew: Renasys GO and Renasys EZ Plus to be used with the Renassys-F/P and Renassys-G Use of the medical devices and applicable consumption items according to manufacturers guidelines and FDA regulations.
  Other Names: Vacuum assisted closure; Vacuum assisted wound closure
  Arms: Negative Pressure Wound Therapy
Other: Standard Wound Therapy — Standard wound therapy according to current evidence-based guideline (basic and advanced methods of wound treatment)
  Other Names: Standard Conventional Wound Therapy
  Arms: Standard Conventional Wound Therapy

SUMMARY:
The purpose of this study is to determine whether Negative Pressure Wound Therapy (NPWT) or Standard Conventional Wound Therapy (SCWT) are effective in the treatment of Iatrogenic Subcutaneous Abdominal Wound healing-impairments (ISAW).

DETAILED DESCRIPTION:
The aim of the study is the comparison between NPWT and Standard Conventional Wound Therapy (SCWT) under clinical, safety and economic aspects in the treatment of postoperative Iatrogenic Subcutaneous Abdominal Wounds (ISAW). The hypothesis is based on the assumption that the application of NPWT for the treatment of postoperative abdominal wound healing impairments (with intact fascia) results in a decrease of time until achievement of wound closure (with confirmation after 30 consecutive days) and for this reason more wound closures can be achieved in the maximum treatment period of 42 days compared to the control therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute subcutaneous abdominal wound-healing impairment after surgical intervention
* Sizes of wound opening (maximum diameter ≥ 3 cm)
* Wound surface ≥ 9 qcm

Exclusion Criteria:

Lack of infrastructure for outpatient continuation of treatment and study-specific interventions

* Existence of an open abdominal fascia
* Acute serious organ failure
* Application of an other active vacuum device at the wound treated during the study conduct within 8 days before screening visit
* Ongoing / during 3 weeks after chemo therapy
* Ongoing / during 3 weeks after radiation therapy Contraindications in accordance with the safety precautions issued by the FDA or the companies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Wound closure | within 42 days of treatment
  Time-of-closure (in days) achieved and confirmed wound closures and rate-of-closure (in number). The wound closure is defined as 100% epithelialization; no need for drainage, no need for supportive therapy or a means of assistance and absence of suture material.
  The closure must remain at least for a period of 30 days.

SECONDARY OUTCOMES:
Wound volume | within the observation period of 180 days
  Reduction of wound volume (cubic centimeter) in the course of treatment.
Wound infections | within the observation period of 180 days
  Number of wound infections over the time.
Recurrences | wthin observation period of 180 days
  Number of recurrences over the time.
Pain | within a maximum treatment time of 42 days
Quality of Life | within observation period of 180 days
  EQ-5D at inclusion, end of maximum treatment time or end of therapy, Follow-Up after 180 days.
Direct costs | within a maximum treatment time of 42 days or until end of therapy
  direct medical resource use and costs: hospitalization, outpatient contact with study centre and other providers, reimbursable drugs, medical sundries, adjuvants, reimbursable services direct non-medical resource use and costs: services, travel costs, expenditure of time for patients, expenditure of time for lay care
Indirect costs | within a maximum treatment time of 42 days or until end of therapy
  Disability, disability pension, premature death
Serious adverse events | within the observation period of 180 days
Adverse events | within a maximum treatment time of 42 days
  Wound- and device-specific adverse events

CONTACTS AND LOCATIONS:
Locations (34):
- Germany (34):
  - Krankenhaus Martha-Maria Halle-Dölau, Halle, Saxony-Anhalt
  - St. Marien-Krankenhaus Ahaus-Vrede, Ahaus
  - Asklepios Stadtklinik Bad Tölz GmbH, Bad Tölz
  - Bundeswehrkrankenhaus Berlin, Berlin
  - Klinikum Bilefeld - Mitte, Bielefeld
  - Knappschaftskrankenhaus Bochum der Ruhr, Bochum
  - Klinikum Darmstadt, Chirurgische Klinik III, Darmstadt
  - Diakonissenkrankenhaus Dessau /Roßlau, Dessau
  - Krankenhaus Düren gem. GmbH, Düren
  - Klinik für Gefäß- und Endovascular-Chirurgie, Klinikum der Johann Wolfgang Goethe - Universität, Frankfurt am Main
  - Krankenhaus St. Elisabeth und St. Barbara, Klinik für Allgmein- und Visceralchirurgie, Halle
  - Universitätsklinikum Halle/Saale, Allgemein-, Viszeral- und Gefäßchirurgie, Halle
  - Asklepios Westklinikum Hamburg, Hamburg
  - Sana Klinikum Hameln-Pyrmont Klinik für Allgemein- und Visceralchirurgie, Hamelin
  - Gemeinschaftskrankenhaus Herdecke, Herdecke
  - Universitätsklinikum Jena, Klinik für Allgemein-, Viszeral- und Gefäßchirurgie, Jena
  - Universitätsklinikum Jena, Klinik für Frauenheilkunde und Geburtshilfe, Abt. Gynäkologie, Jena
  - Westpfalz-Klinikum GmbH, Klinikum für Allgemein-, Viszeral- und Transplantationschirurgie, Kaiserslautern
  - Städtisches Klinikum Karlsruhe gGmbH, Klinik für Allgemein- und Viszeralchirurgie, Karlsruhe
  - Kliniken der Stadt Köln Krankenhaus Merheim, Klinik für Visceral-, Gefäß- und Transplantationschirurgie, Köln-Merheim
  - Universitätsklinikum Schleswig-Holstein, Klinik für Chirurgie, Lübeck
  - Klinik und Poliklinik für Allgemein- und Abdominalchirurgie, Johannes Gutenberg- Universität, Mainz
  - Wundzentrum München, München
  - Klinikum der Universität München, Chirurgische Klinik und Poliklinik, München-Großhadern
  - Universitätsklinikum Münster, Klinik für Allgemein und Viszeralchirurgie, Münster
  - Städtisches Klinikum Neunkirchen, Neunkirchen/Saar
  - Ortenauklinikum Offenburg-Gengenbach, Offenburg
  - Klinikum Dorothea Christiane Erxleben, Quedlinburg
  - Carl-von-Basedow Klinikum, Saalekreis, Querfurt
  - Zentrum für Gefäßmedizin Klinikum Südstadt Rostock, Rostock
  - Asklepios Klinikum Uckermark GmbH, Klinik für Allgemein- und Visceralchirurgie, Schwedt
  - Agaplesion Bethesda-Krankenhaus Stuttgart, Stuttgart
  - HSK Dr. Horst Schmidt Kliniken, Wiesbaden
  - Evangelisches Krankenhaus Paul Gerhardt Stift, Allgemein-, Viszeral- und Gefäßchirurgie, Wittenberg